CLINICAL TRIAL: NCT06458530
Title: Vivo Prediabetes Study: Evaluating the Effect of Participating in Vivo on Physical Function and Glycemic Level in Sedentary Older With Prediabetes
Brief Title: Examining the Effects of Vivo on Physical Function and Glycemic Level in Sedentary Older With Prediabetes.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Impactiv, Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Eric Levian, CEO, Impactiv, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00110021_2
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: PreDiabetes; Older Adult; Muscle Loss; Muscle Weakness
Keywords: Virtual Exercise Intervention; Strength training; Older Adult; Prediabetes; Muscle strength; Small group training
MeSH Terms: conditions — Prediabetic State; Muscular Atrophy; Muscle Weakness

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The PI will be masked to randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vivo intervention (Experimental): Participants will meet virtually twice a week for 12 weeks with their small group and certified trainer for 45 minutes.
  Interventions: Behavioral: Vivo
- Waitlist control (No Intervention): Participants randomized to this arm will be asked to maintain their baseline physical activity for 12-weeks. They will be scheduled for the baseline and 12-week assessment and following the 12-week assessment, they will be offered enrollment into Vivo.

INTERVENTIONS:
Behavioral: Vivo — Participants will meet virtually twice a week with their small group and certified trainer for 45 minutes exercise sessions for a 12-week period.
  Arms: Vivo intervention

SUMMARY:
This is a 12-week randomized, controlled trial that seeks to examine the effect of Vivo on 1) change in lower extremity strength defined as number of chair stands done in 30 seconds and 2) change in average glycemic level (HbA1c) compared to a wait list control.

DETAILED DESCRIPTION:
This is a 12-week randomized, controlled trial that seeks to examine the effect of Vivo on 1) change in lower extremity strength defined as number of chair stands done in 30 seconds and 2) change in average glycemic level (HbA1c) compared to a wait list control. After informed consent and baseline assessments, up to 90 individuals will be randomized in one of two arms: 1) Vivo intervention or 2) waitlist control. Participants in the Vivo 2.0 intervention arm will meet virtually twice a week with their small group and certified trainer for 45 minutes over a 12-week period. Participants will be men and women, ≥60 years old, sedentary, with prediabetes and low function. All participants will undergo baseline and 12-week assessments

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Ambulatory and community-dwelling
* Diagnosis of Pre-diabetes within prior 12 months: fasting glucose between 100 to 126 OR HbA1c between 5.7 and 6.4%
* Low functioning: 1) able to do at least 1 chair stand and 2) number of chair stands done in 30 seconds is below criterion-referenced fitness standards for maintaining physical independence for age and gender
* Sedentary: less than 150 minutes of moderate physical activity OR less than 60 minutes of vigorous physical activity per week
* Have not engaged in resistance training for at least 6 months prior to enrollment
* Access to WiFi in defined exercise space

Exclusion Criteria:

* Inability to complete physical function assessment
* Use of antidiabetic medications
* Use of testosterone supplement or replacement
* Clinical disorder precluding/interfering with participation of assessments

  * Unstable angina, arrhythmia, uncontrolled hypertension
  * End Stage Renal Disease on Hemodialysis
  * Lower extremity amputation or paralysis
  * Neurological condition causing functional or pronounced cognitive impairments
  * Active malignancy except for non-melanomatous skin cancers
* Weight instability (defined as gain or loss of ≥10% over the last 6 months)
* Unable to provide consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Lower body strength | baseline and 12 weeks
  Lower body strength measured by the 30-second chair stand

SECONDARY OUTCOMES:
Hemoglobin A1C (HbA1C) | baseline and 12 weeks
  Hemoglobin A1C (HbA1C) measure during clinic assessment
Balance | baseline and 12 weeks
  Static Balance Score of the SPPB. Sore 0-4 depending on the combined results of side by side, semi-tandem, and tandem stand tests.
Physical Activity Level | baseline and 12 weeks
  Average step count using Garmin Fitness Tracker
Aerobic Endurance | baseline and 12 weeks
  Measured by the 2-minute step test for aerobic endurance

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No